CLINICAL TRIAL: NCT05155891
Title: Prospective, Non-Randomized, Controlled Investigation of Prostate Artery Embolization Compared to Holmium Laser Enucleation of Prostate for the Treatment of Symptomatic Benign Prostatic Hyperplasia in Prostate Glands Larger Than 80 Grams
Brief Title: Investigation of Prostate Artery Embolization Compared to Holmium Laser Enucleation of Prostate
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Hemendra Shah, Professor of Clinical Urology, University of Miami
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20210029
Record Dates: First submitted 2021-11-30; First posted 2021-12-14 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-05

CONDITIONS: Benign Prostatic Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Embosphere Microspheres group (Experimental): Participants in this group who are undergoing standard of care (SOC) prostate artery embolization (PAE) for treatment of their symptomatic benign prostatic hyperplasia (BPH) will receive Embosphere Microspheres during scheduled SOC PAE surgery.
  Interventions: Device: Embosphere Microspheres
- HoLEP Group (Active Comparator): Participants in this group who are undergoing SOC PAE for treatment of their symptomatic benign prostatic hyperplasia (BPH) will receive SOC Holmium laser enucleation of prostate (HoLEP).
  Interventions: Procedure: HoLEP Procedure

INTERVENTIONS:
Device: Embosphere Microspheres — The SOC PAE procedure will be performed by attempting to embolize prostatic arteries of both sides in a single session with 300-500 um Embosphere Microspheres. The microspheres will be mixed with a contrast agent and will be delivered to the arteries supplying the prostate via a microcatheter.
  Arms: Embosphere Microspheres group
Procedure: HoLEP Procedure — The SOC PAE procedure will be performed with the SOC HoLEP as per standard institutional guidelines. The HoLEP procedure involves passing a telescope through the urethra and removing the central part of the prostate gland using a laser.
  Arms: HoLEP Group

SUMMARY:
The purpose of this research study is to evaluate prostate artery embolization (PAE) compared to Holmium laser enucleation of prostate (HoLEP) in improving a patient's overall prostate related symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is age 50 or older.
2. Patient has signed informed consent and agrees to attend all follow-up study visits.
3. Patient has had LUTS secondary to BPH or any complications secondary to BPH and qualifying for active intervention.
4. Patient has a baseline IPSS Score > 13 at baseline.
5. Patient has a prostate size of at least 80 grams and not more than 250 grams, measured by magnetic resonance imaging (MRI) or transrectal ultrasonography (TRUS).
6. Patient has BPH symptoms refractory to medical treatment or for whom medication is contraindicated, not tolerated, or refused.
7. Patient must be a candidate for HoLEP or PAE.

Exclusion Criteria:

1. Subject has untreated active infection (e.g., active urinary tract infection or prostatitis)
2. Subject has a diagnosis or received treatment for chronic prostatitis or chronic pelvic pain syndrome (e.g., nonbacterial chronic prostatitis).
3. Patients with indwelling urinary catheters or those performing self-catheterization.
4. Biopsy proven prostate or bladder cancer.

   - Patient with elevated PSA will be counselled by urologist and a shared decision will be made with the patient after discussion about pros and cons of prostate biopsy.
5. Patients with neurogenic bladder disorder.
6. Urethral stricture, bladder neck contracture, sphincter abnormalities, urinary obstruction due to causes other than BPH, or other potentially confounding bladder or urethral disease or condition.
7. Patients with prior history transurethral resection of the prostate (TURP), Green Light laser treatment, or other prostate surgical treatments within past year(12 months).
8. Any known condition that limits catheter-based intervention or is a contraindication to embolization, such as intolerance to a vessel occlusion procedure or severe atherosclerosis.
9. Cardiac condition including congestive heart failure or arrhythmia, uncontrolled diabetes mellitus, significant respiratory disease or known immunosuppression which required hospitalization within the previous 6 months.
10. Acute myocardial infarction, open heart surgery, or cardiac arrest within 180 days prior to the date of informed consent.
11. Patient is interested in future fertility and wish to preserve ejaculation will be excluded from HoLEP arm
12. History of coagulation cascade disorders (which are not normalized by medical treatment before the procedure) or disorders that affect platelet count or function (e.g., von Willebrand disease) that would put the subject at risk for intraoperative or postoperative bleeding.
13. History of major allergic reaction to iodinated contrast agents will be excluded from PAE arm.
14. History of hypersensitivity to gelatin products will be excluded from PAE arm.
15. Subject has a life expectancy of less than 2 yrs.
16. Post void residual more than 500 ml at baseline.
17. Participation in any other BPH trials during the time of study.

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2022-06-17 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Change in BPH symptoms as measured by the IPSS | Baseline, 3 months
  The International Prostate Symptom Score (IPSS) has a total score ranging from 0-35 with the higher score indicating more severe symptoms

SECONDARY OUTCOMES:
Duration of hospitalization after the procedure | up to 48 hours
  The duration of hospitalization associated with each procedure will be calculated in hours.
Duration of urinary catheterization after the procedure | up to 48 hours
  The duration of urinary catheterization associated with each procedure will be calculated in hours.
Change in BPH symptoms as measured by IPSS | Baseline, 12 months
  International Prostate Symptom Score (IPSS) has a total score ranging from 0-35 with the higher score indicating more severe symptoms
Change in peak urine flow rate | Baseline, 12 months
  The peak urine flow rate (Qmax) will be measured via uroflowmetry
Change in post-void residual urinary volume (PVR) | Baseline, 12 months
  PVR will be measured using an ultrasound bladder scanner
Change in erectile function as measured by the IIEF | Baseline, 12 Months
  The International Index of Erectile Function (IIEF) has a total score ranging from 0-25 with higher score indicating better erectile function
Change in retrograde ejaculation as measured by the Ejaculatory questionnaire | Baseline, 12 Months
  The Ejaculatory Questionnaire has a total score ranging from 0-20 with the higher score indicating better outcomes
Change in incontinence as measured by the ICIQ - UI SF | Baseline, 12 Months
  The International Consultation on Incontinence Questionnaire (ICIQ) -Urinary Incontinence (UI) Short Form (SF) is a 4-item self-report of urinary incontinence to document changes in bladder function. Scores range from 0-21, with greater values indicating increased severity.
Change in mean prostate volume | Baseline, 12 months
  As measured by Magnetic Resonance Imaging (MRI) and transrectal ultrasound (TRUS)
Change in prostate specific antigen (PSA) levels | Baseline, 12 Months
  As measured by serum blood samples
Incidence of adverse events | Up to 12 Months
  As evaluated by treating physician
Incidence of procedure-related adverse events | Up to 12 Months
  As evaluated by treating physician
Change in medication use related to BPH-LUTS | Baseline, 12 Months
  Change in BPH lower urinary tract symptoms (LUTS) medication use (including alpha blockers, 5-alpha reductase inhibitors and phosphodiesterase type 5 (PDE5) inhibitors) will be reported

CONTACTS AND LOCATIONS:
Overall Officials: Hemendra Shah, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No